CLINICAL TRIAL: NCT00942084
Title: An Open Label Study to Describe the Pharmacokinetics of Acyclovir in Premature Infants
Brief Title: A Study to Describe the Pharmacokinetics of Acyclovir in Premature Infants (PTN_Acyclo)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phillip Brian Smith (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Phillip Brian Smith, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00028772
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Herpes Simplex Virus; Neonatal Sepsis
Keywords: HSV; Acyclovir; Pharmacokinetics; Neonate; Premature; Sepsis
MeSH Terms: conditions — Herpes Simplex; Neonatal Sepsis; Premature Birth; Sepsis | interventions — Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Protocol V2&up-Grp1-Acyclo10 mg/kg IVq12 (Active Comparator): Gestational Age 23-29 weeks Postnatal Age < 14 days Dosage 10 mg/kg IV q12 Number of Infants 8
  Interventions: Drug: Acyclovir
- Protocol V2&up-Grp2_Acyclo20 mg/kg IVq12 (Active Comparator): Gestational Age 23-29 weeks Postnatal Age 14-44 days Dosage 20 mg/kg IV q12 Number of Infants 8
  Interventions: Drug: Acyclovir
- Protocol V2&up-Grp3-Acyclo20 mg/kg IVq8 (Active Comparator): Gestational Age 30-34 weeks Postnatal Age <45 days Dosage 20 mg/kg IV q8 Number of Infants 4
  Interventions: Drug: Acyclovir
- Protocol V1-Grps1-4-Acyclo 500 mg/m2 IVq8h (Other): All patients in protocol V1 were to be dosed with 500 mg/m2 IV q8h. Protocol V1 Group 1: Gestational Age: 23-29 Weeks; PNA: <14 days; Protocol V1 Group 2: Gestational Age: 30-42 Weeks; PNA: <14 days; Protocol V1 Group 3: Gestational Age: 23-29 Weeks; PNA: 14-60 days; Protocol V1 Group 4: Gestational Age: 30-42 Weeks; PNA: 14-60 days
  Interventions: Drug: Acyclovir

INTERVENTIONS:
Drug: Acyclovir — Protocol V2 & up: Acyclovir 7mg/ml to be administered IV at 10 mg/kg IV q12 or 20 mg/kg IV q12 or 20 mg/kg IV q8 for a total of 6-9 doses(3 days).
  Protocol V1: Acyclovir 5 mg/mL to be administered IV at 500 mg/m2 IV q8h for a total of approximately 15 doses (10 days).

SUMMARY:
Acyclovir is a drug used to treat herpes simplex virus (HSV) infections in babies. Appropriate dosing of acyclovir is known for adults and children but acyclovir has not been adequately studied in full-term or premature neonates. HSV is a very serious infection in babies <6 months of age and often results in death or profound mental retardation. HSV leads to profound mental retardation in young infants because the virus attacks the central nervous system.

The investigators hypothesize that the currently recommended dose of acyclovir is inadequate to produce adequate blood levels to combat herpes simplex infection. The investigators propose to study acyclovir levels in the blood of babies who are placed on acyclovir to treat a suspected HSV infection. This will allow them to determine the appropriate dose in premature infants. This is an unmet public health need because it is likely that the drug behaves differently in premature infants than it does in term infants and older children. Premature babies have more body water and less body tissue. Their kidneys are more immature and do not function as well as full term infants. Premature neonates are also at the greatest risk from herpes infection because they have poorly functioning immature immune systems. Early and appropriate treatment with acyclovir has resulted in improved outcome in term infants.

DETAILED DESCRIPTION:
Neonatal herpes infection carries a major risk of death if untreated. Prognosis is related to disease extent and timing of therapy, making early diagnosis crucial. Mortality in the pre-antiviral era was 90% for disseminated disease and 50% for central nervous system (CNS) disease. Institution of high-dose (60 mg/kg/day) antiviral therapy with acyclovir has reduced mortality to 31% for disseminated disease and 6% for CNS disease.1 Although acyclovir has reduced mortality dramatically, morbidity remains high.

Study population: Infants < 45 days postnatal age, suspected to have a systemic infection divided into groups by gestational and postnatal age:

Group-1: 23-29 weeks gestational age, <14 days postnatal age Group-2: 23-29 weeks gestational age, 14-44 days postnatal age Group-3: 30-34 weeks gestational age, <45 days postnatal age

Intravenous acyclovir will be administered for 3 days.

Timing of PK sample collection will be with respect to the end of each IV infusion. Timed PK sampling will be drawn at doses 1, and doses 5, 6, 7, 8, or 9.

Dose 1:

0-15 minutes after completion of the 1st dose; Within 30 minutes prior to administration of 2nd dose

Steady state [doses 5 or 6 (groups 1 and 2), doses 8 or 9 (group 3)]:

Within 30 minutes prior to dose; 0-15 minutes after completion of the dose; 2-3 hours after completion of the dose; Within 30 minutes prior to administration of the next dose

Last dose:

6-7 hours after the last dose (groups 1 and 2)and 10-11 hours after the last dose (group 3)

ELIGIBILITY:
The investigator or other study site personnel will document in the source documents (e.g., the hospital chart) that informed consent was obtained. Laboratory tests or non-pharmacologic treatment procedures that were performed as standard of care within 72 hours prior to first dose of study drug may be used for screening procedures and recorded in the CRF.

Inclusion Criteria

1. < 45 days of age at the time of initial study drug administration.
2. Sufficient venous access to permit administration of study medication.
3. Availability and willingness of the parent/legal guardian to provide written informed consent.
4. Suspected HSV sepsis OR At least two (2) of the following

   * Signs of sepsis AND negative blood cultures for >24 hours7
   * Respiratory distress8
   * Lethargy8
   * Fever ≥ 38.0°C7
   * Skin lesions7,8
   * Seizures (clinical OR EEG confirmed)7
   * Irritability7
   * AST OR ALT >2 X upper limit of normal7,8
   * >20 WBCs/µL or >500 RBCs/µL7

Exclusion Criteria

1. History of anaphylaxis attributed to acyclovir.
2. Serum creatinine >1.7 mg/dL.
3. Urine output <0.5 mL/kg/hour over the previous 12 hours
4. Previous participation in the study.
5. Concomitant condition, which in the opinion of the investigator would preclude a participant's participation in the study

Max Age: 45 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip B Smith, M.D., Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Wesely Medical Center, Wichita, Kansas
  - Tulane School of Medicine, New Orleans, Louisiana
  - Duke University, Durham, North Carolina

REFERENCES:
- [Background] Whitley RJ. Herpes simplex virus infection. Semin Pediatr Infect Dis. 2002 Jan;13(1):6-11. doi: 10.1053/spid.2002.29752. PMID 12118847
- [Background] Kimberlin DW, Lin CY, Jacobs RF, Powell DA, Corey L, Gruber WC, Rathore M, Bradley JS, Diaz PS, Kumar M, Arvin AM, Gutierrez K, Shelton M, Weiner LB, Sleasman JW, de Sierra TM, Weller S, Soong SJ, Kiell J, Lakeman FD, Whitley RJ; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. Safety and efficacy of high-dose intravenous acyclovir in the management of neonatal herpes simplex virus infections. Pediatrics. 2001 Aug;108(2):230-8. doi: 10.1542/peds.108.2.230. PMID 11483782
- [Background] Lietman PS. Acyclovir clinical pharmacology. An overview. Am J Med. 1982 Jul 20;73(1A):193-6. doi: 10.1016/0002-9343(82)90089-4. PMID 7048912
- [Background] Englund JA, Fletcher CV, Balfour HH Jr. Acyclovir therapy in neonates. J Pediatr. 1991 Jul;119(1 Pt 1):129-35. doi: 10.1016/s0022-3476(05)81053-4. PMID 2066845
- [Background] Blum MR, Liao SH, de Miranda P. Overview of acyclovir pharmacokinetic disposition in adults and children. Am J Med. 1982 Jul 20;73(1A):186-92. doi: 10.1016/0002-9343(82)90088-2. PMID 7048911
- [Background] Hintz M, Connor JD, Spector SA, Blum MR, Keeney RE, Yeager AS. Neonatal acyclovir pharmacokinetics in patients with herpes virus infections. Am J Med. 1982 Jul 20;73(1A):210-4. doi: 10.1016/0002-9343(82)90093-6. PMID 6285713
- [Background] Yeager AS. Use of acyclovir in premature and term neonates. Am J Med. 1982 Jul 20;73(1A):205-9. doi: 10.1016/0002-9343(82)90092-4. PMID 6285712
- [Background] Pickering LK. Red Book. 28th ed. Elk Grove Village, Illinois: American Academy of Pediatrics; 2009.
- [Background] Kimberlin DW. When should you initiate acyclovir therapy in a neonate? J Pediatr. 2008 Aug;153(2):155-6. doi: 10.1016/j.jpeds.2008.04.027. No abstract available. PMID 18639724
- [Background] Brigden D, Bye A, Fowle AS, Rogers H. Human pharmacokinetics of acyclovir (an antiviral agent) following rapid intravenous injection. J Antimicrob Chemother. 1981 Apr;7(4):399-404. doi: 10.1093/jac/7.4.399. No abstract available. PMID 7251524
- [Background] Feldman S, Rodman J, Gregory B. Excessive serum concentrations of acyclovir and neurotoxicity. J Infect Dis. 1988 Feb;157(2):385-8. doi: 10.1093/infdis/157.2.385. No abstract available. PMID 3335815
- [Result] Rhodin MM, Anderson BJ, Peters AM, Coulthard MG, Wilkins B, Cole M, Chatelut E, Grubb A, Veal GJ, Keir MJ, Holford NH. Human renal function maturation: a quantitative description using weight and postmenstrual age. Pediatr Nephrol. 2009 Jan;24(1):67-76. doi: 10.1007/s00467-008-0997-5. Epub 2008 Oct 10. PMID 18846389

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total enrollment is 32. 32 for safety analysis and 30 in PK population (28 included in final PK analysis).
Groups:
- Acyclovir Study Enrollment: Two open-label PK studies contributed the data for this report. Version 1 was single-center and Version >=2 was multi-center. Acyclovir was administered intravenously as a 1-hour infusion for up to 3 days. Dosing in Study 1 was 500 mg/m2 every 8 hours. Dosing in Study 2 was determined by GA and PNA: 10 mg/kg every 12 hours (23-29 weeks GA and <14 days PNA); 20 mg/kg every 12 hours (23-29 weeks GA and 14-44 days PNA); and 20 mg/kg every 8 hours (30-34 weeks GA and <45 days PNA).
Period: Overall Study
Arm/Group | Acyclovir Study Enrollment
Started | 32
Completed | 30 (There were 2 infant deaths. None determined to be related to study drug.)
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Groups:
- Acyclovir Study Design: Two open-label PK studies contributed the data for this report. Version 1 was single-center and Version >=2 was multi-center. Acyclovir was administered intravenously as a 1-hour infusion for up to 3 days. Dosing in Study 1 was 500 mg/m2 every 8 hours. Dosing in Study 2 was determined by GA and PNA: 10 mg/kg every 12 hours (23-29 weeks GA and <14 days PNA); 20 mg/kg every 12 hours (23-29 weeks GA and 14-44 days PNA); and 20 mg/kg every 8 hours (30-34 weeks GA and <45 days PNA).
Arm/Group | Acyclovir Study Design
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: days]
  Postnatal Age (days) | 3.0 [0.0 to 30.0]
Age, Continuous [Median (Full Range); unit: weeks]
  Gestational Age (weeks) | 30.5 [23.0 to 40.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32
Birthweight [Median (Full Range); unit: grams] | 1295 [420 to 4840]

OUTCOME MEASURES:

1. Primary Outcome: Clearance (CL)
Description: Timeframe:
  Version 1:0-5 min,2-4 hrs,6-8 hrs post doses 1 and 5-15; prior to doses 5-15 Version 2:0-15 min post doses 1 and 5-15; within 30 min prior to doses 2 and 5-15; 2-3 hrs post doses 5-15; 15-18 hrs post last dose
Time Frame: V1:0-5 min,2-4 hrs,6-8 hrs post Doses 1&5-15;prior to doses 5-15; V2:0-15 min post doses 1&5-15; within 30 min prior to doses 2&5-15; 2-3 hrs post doses 5-15; 15-18 hrs post last dose
Population: 32 infants enrolled. 2 infants died. 2 infants did not contribute PK samples to the analysis. 28 contributed PK samples to the final analysis.
Measure: Median (Full Range); unit: L/h/kg
Arm/Group | Acyclovir Study Design
Number analyzed (Participants) | 28
L/h/kg | 0.278 [0.095 to 0.812]

2. Primary Outcome: Volume of Distribution (V)
Time Frame: up to 3 days of study drug administration and 10 days of safety monitoring
Population: as for outcome 1
Measure: Median (Full Range); unit: L/kg
Arm/Group | Acyclovir Study Design
Number analyzed (Participants) | 28
L/kg | 3.34 [0.293 to 10.85]

3. Primary Outcome: Half-life (T1/2)
Time Frame: up to 3 days of study drug administration and 10 days of safety monitoring
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Acyclovir Study Design
Number analyzed (Participants) | 28
h | 7.07 [1.61 to 13.2]

4. Primary Outcome: Maximum Steady State Concentration (Cmaxss)
Time Frame: up to 3 dasy of study drug administration and 10 days of safety monitoring
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/L
Arm/Group | Acyclovir Study Design
Number analyzed (Participants) | 28
mg/L | 11.1 [4.59 to 110]

5. Primary Outcome: Steady State Concentration at 50% of the Dosing Interval (C50ss)
Time Frame: up to 3 days of study drug administration and 10 days of safety monitoring
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/L
Arm/Group | Acyclovir Study Design
Number analyzed (Participants) | 28
mg/L | 6.33 [3.38 to 65.7]

6. Primary Outcome: Minimum Steady State Concentration (Cminss)
Time Frame: up to 3 days of study drug administration and 10 days of safety monitoring
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/L
Arm/Group | Acyclovir Study Design
Number analyzed (Participants) | 28
mg/L | 4.15 [2.19 to 39.3]

ADVERSE EVENTS:
Time Frame: Up to 3 days of study drug administration and 10 days of safety monitoring
Arm/Group | Acyclovir Study Design
Serious Adverse Events (participants affected / at risk) | 4/32
Other Adverse Events (participants affected / at risk) | 21/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir Study Design (N=32)
Death (General disorders) | 2 (2) — 1 infant died due to nonketotic hyperglycinaemia and 1 infant dies due to sepsis.
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyclovir Study Design (N=32)
Haemolytic anemia (Blood and lymphatic system disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Congenital cardiovascular anomaly (Congenital, familial and genetic disorders) | 7 (7)
Nonketotic hyperglycinaemia (Congenital, familial and genetic disorders) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 3 (3)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Blood creatinine abnormal (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Neonatal hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infantile apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No